CLINICAL TRIAL: NCT05617352
Title: The Impact of Two-field or Three-field Lymphadenectomy on Overall Survival in Middle and Lower Thoracic Esophageal Squamous Cell Carcinoma: A Single Center Retrospective Analysis
Brief Title: The Impact of Two-field or Three-field Lymphadenectomy on Overall Survival in Middle and Lower Thoracic Esophageal Squamous Cell Carcinoma: An Observational Study
Status: Completed | Type: Observational
Sponsor: Yongtao Han (Other)
Responsible Party: Sponsor-Investigator, Yongtao Han, Clinical Professor, Sichuan Cancer Hospital and Research Institute
Organization: Sichuan Cancer Hospital and Research Institute (Other)
Other Study IDs: SCCH-TS2204
Record Dates: First submitted 2022-11-07; First posted 2022-11-15 (Actual); Last update posted 2022-11-21 (Actual); Status verified 2022-11

CONDITIONS: Esophageal Cancer
MeSH Terms: conditions — Esophageal Neoplasms

STUDY DESIGN:
Observational Model: Other | Time Perspective: Retrospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- 2F Group: Patients with Two-field Lymphadenectomy
  Interventions: Diagnostic Test: Since the data were collected retrospectively, there were no interventions
- 3F Group: Patients with Three-field Lymphadenectomy
  Interventions: Diagnostic Test: Since the data were collected retrospectively, there were no interventions

INTERVENTIONS:
Diagnostic Test: Since the data were collected retrospectively, there were no interventions — Since the data were collected retrospectively, there were no interventions

SUMMARY:
To clarify the effect of Two-field or Three-field Lymphadenectomy on the survival of esophageal squamous cell carcinoma.

ELIGIBILITY:
Inclusion Criteria:

* 1. Men and women aged 18-85 years
* 2. Histologically confirmed primary thoracic esophageal squamous cell carcinoma,
* 3. Staging PT1b-4A, N0-3, M0 AJCC eighth edition
* 4. Excluding lymph node dissection < 15, (meeting the guideline criteria)
* 5. The tumor located in the lower middle thoracic.

Exclusion Criteria:

* 1. Patients with a history of previous thoracic and abdominal surgery that may affect lymphatic reflux
* 2. Patients with distant metastasis confirmed by imaging
* 3. Patients with obvious surgical contraindications.

Ages: 18 Years to 90 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients with esophageal cancer and need surgical treatment.
Sampling Method: Non-Probability Sample
Enrollment: 1659 (Actual)
Dates: Start 2022-05-01 (Actual); Primary Completion 2022-10-01 (Actual); Study Completion 2022-10-10 (Actual)

PRIMARY OUTCOMES:
The number of lymph nodes | 2010.1.1-2017.12.30
  Surgical data were retrospectively collected

CONTACTS AND LOCATIONS:
Locations (1):
- Sichuan Cancer Hospital, Chengdu, Sichuan, China

IPD SHARING:
Plan to Share IPD: Undecided
We are willing to share data, analytic methods, and study materials related to this article with other researchers. Provided that all of the above will not be used for commercial or profit purposes. Other researchers can contact the corresponding author of this article by email and indicate the required research materials and purpose. We will be glad to provide relevant materials for this study after approval and discussion.